CLINICAL TRIAL: NCT00302016
Title: An Open-label, Multicenter, Expanded Access Study of Oral AMN107 in Adult Patients With Imatinib-resistant or Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase, or Chronic Phase.
Brief Title: Expanded Access Program of AMN107 in Imatinib-resistant or Intolerant Adult Patients With Chronic Myeloid Leukemia
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107A2109; NCT00532649 (obsolete NCT alias)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; AMN 107; Imatinib resistant or intolerant; nilotinib; enact
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

INTERVENTIONS:
Drug: AMN107

SUMMARY:
This study will further evaluate if AMN107 is safe in adults with chronic myeloid leukemia who are resistant or intolerant to imatinib and to provide patients access to this new drug until the drug becomes commercially available.

ELIGIBILITY:
Inclusion criteria:

* Imatinib-resistant or -intolerant Philadelphia chromosome-positive chronic myeloid leukemia in blast crisis, accelerated phase, or chronic phase.
* Chronic myeloid leukemia patients who have been treated with an investigational tyrosine kinase inhibitor.
* Laboratory values within normal limits.

Exclusion criteria:

* Impaired cardiac function.
* Acute or chronic liver or renal disease considered unrelated to tumor.
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients who are currently receiving treatment with any of the medications that have the potential to prolong the QT interval or to inhibit the metabolism of AMN107 (CYP3A4/5 inhibitors).
* Patients with a history of another malignancy that is currently clinically significant or currently requires active intervention.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (270):
- United States (59):
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center-Lombardi Cancer Center, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Osler Medical Inc./Osler Clinical Research, Melbourne, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Integrated Community, Orange Park, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - MD Anderson Cancer Center, Orlando, Florida
  - Hematology Oncology Assoc., Pensacola, Florida
  - Emory University Cancer Institute, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Stroger Cook County Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital & Health Centers, Beech Grove, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Louisville Oncology Research, Louisville, Kentucky
  - LSU Health Sciences Center, Shreveport, Louisiana
  - St. Agnes Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - St. John Hospital and Medical Center, Grosse Pointe, Michigan
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Cancer Institute of New Mexico, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop Hematology/Oncology, Mineola, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Three Medical Park, Columbia, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington
- Novartis Investigative Site, Saint Leonards, Australia
- Austria (5):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Wels
- Belgium (14):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Arlon
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Yvoir
- Brazil (9):
  - Novartis Investigative Site, Belo Horizonte
  - Novartis Investigative Site, Brasilia-DF
  - Novartis Investigative Site, Campinas
  - Novartis Investigative Site, Curitaba
  - Novartis Investigative Site, Curitiba
  - Novartis Investigative Site, Porto Alegre-RS
  - Novartis Investigative Site, Ribeirão Preto
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Canada (7):
  - Novartis Investigative Site, Edmonton
  - Novartis Investigative Site, Halifax
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Ottawa
  - Novartis Investigative Site, Toronto
  - Novartis Investigative Site, Vancouver
- China (4):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjing
- Czechia (5):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Plzen-Lochotin
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Vejle
- France (22):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (30):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Pokfulam, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Dublin, Ireland
- Italy (36):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Bolzano
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Campobasso
  - Novartis Investigative Site, Catania
  - Novartis Investigative Site, Catanzaro
  - Novartis Investigative Site, Ferrara
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Nuoro
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Perugia
  - Novartis Investigative Site, Pesaro
  - Novartis Investigative Site, Pescara
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Reggio Calabria
  - Novartis Investigative Site, Reggio Emilia
  - Novartis Investigative Site, Rionero in Vulture
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Ronciglione
  - Novartis Investigative Site, San Giovanni Rotundo
  - Novartis Investigative Site, Siena
  - Novartis Investigative Site, Tarante
  - Novartis Investigative Site, Torino
  - Novartis Investigative Site, Udine
  - Novartis Investigative Site, Via Pansini
- Novartis Investigative Site, Beirut, Lebanon
- Malaysia (4):
  - Novartis Investigative Site, Georgetown, Penang
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Pulau Pinang
  - Novartis Investigative Site, Subang Jaya, Selangor
- Novartis Investigative Site, Mexico City, Mexico
- Netherlands (5):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Oslo, Norway
- Poland (5):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
- Russia (6):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Ufa
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Roodepoort, Gauteng
- South Korea (5):
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Deajeon
  - Novartis Investigative Site, Jeollanam-do
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
- Spain (13):
  - Novartis Investigative Site, Baracaldo, Pais Vasco
  - Novartis Investigative Site, Barcelona, Cataluna
  - Novartis Investigative Site, Cataluna
  - Novartis Investigative Site, Granada, Andalucia
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Salamanca, Castilla Y Leon
  - Novartis Investigative Site, San Sabastian, Pais Vasco
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Sweden (5):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Taiwan (5):
  - Novartis Investigative Site, Chiayi City
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Malatya
  - Novartis Investigative Site, Samsun
- United Kingdom (6):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham

REFERENCES:
- [Derived] Zhou L, Meng F, Yin O, Wang J, Wang Y, Wei Y, Hu P, Shen Z. Nilotinib for imatinib-resistant or -intolerant chronic myeloid leukemia in chronic phase, accelerated phase, or blast crisis: a single- and multiple-dose, open-label pharmacokinetic study in Chinese patients. Clin Ther. 2009 Jul;31(7):1568-75. doi: 10.1016/j.clinthera.2009.07.016. PMID 19695406